CLINICAL TRIAL: NCT03937102
Title: Measurement of Cardiac Output in Intensive Care Unit With Unstable Hemodynamic: Validation of Physioflow® Device Versus Trans Thoracic Echocardiography
Acronym: Reacshock
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier de Lens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2018_843_0001
Record Dates: First submitted 2019-04-25; First posted 2019-05-03 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Cardiac Output
Keywords: cardiac output; trans thoracic echocardiography; passive leg raising; volume expansion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cardiac output measure with TTE — All patients included will be simultaneously monitored with transthoracic echocardiography (TTE) and the Physioflow® thoracic electrical bioimpedance device. Cardiac output is measured by the Physioflow® Thoracic Bioimpedance Device and TTE before and after passive leg raising maneuver (PLR)
Procedure: cardiac output measure with Physioflow® thoracic electrical bioimpedance — All patients included will be simultaneously monitored with transthoracic echocardiography (TTE) and the Physioflow® thoracic electrical bioimpedance device. Cardiac output is measured by the Physioflow® Thoracic Bioimpedance Device and TTE before and after passive leg raising maneuver (PLR)

SUMMARY:
Physioflow® is a new device for measuring cardiac output in a non-invasive way using a thoracic bioimpedance technique. This technique has been validated in patients in stress tests as well as in Chronic Obstructive Pulmonary Disease (COPD) patients, in obese patients and in children. Very little work has been published in intensive care unit (ICU) and no studies have been done on hemodynamically unstable patients. The aim of this work is to compare the cardiac output measured by Physioflow® to the transthoracic echocardiography (TTE) in ventilated, sedated patients hospitalized in ICU receiving catecholamines and for whom the attending physician wants to evaluate the fluid responsiveness using the TTE and a passive leg raising maneuver (PLR).

DETAILED DESCRIPTION:
All patients included will be simultaneously monitored with TTE and the Physioflow® thoracic electrical bioimpedance device. Cardiac output is measured by the Physioflow® Thoracic Bioimpedance Device and TTE before and after PLR. If the attending physician decide to administer fluid expansion a new set of cardiac output measurement will be performed before and after the volume expansion.

ELIGIBILITY:
Inclusion Criteria:

* patient more than 18 year-old
* patient sedated and adapted to the assisted controlled ventilation
* patient receiving catecholamine (norepinephrine, epinephrine or dobutamine)
* patient requiring an haemodynamic evaluation by trans-thoracic echocardiography and PLR according to the attending physician

Exclusion Criteria:

* pregnant women
* patients with a poor echogenicity
* patients deprived of public law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient ≥18 year-old, sedated and adapted to the assisted controlled ventilation, receiving catecholamine (norepinephrine, epinephrine or dobutamine), requiring an haemodynamic evaluation by trans-thoracic echocardiography and PLR according to the attending physician.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Measure of cardiac output with transthoracic echocardiography (TTE) before PLR | during one hour , the day of inclusion
  Measure of Cardiac output with transthoracic echocardiography (TTE) before passive leg raising maneuver (PLR)
Measure of Cardiac output with Physioflow before PLR | during one hour , the day of inclusion
  Measure of Cardiac output with Physioflow before passive leg raising maneuver (PLR)
Measure of cardiac output with transthoracic echocardiography (TTE) after PLR | during one hour , the day of inclusion
  Measure of cardiac output with transthoracic echocardiography (TTE) after passive leg raising maneuver (PLR)
Measure of cardiac output with Physioflow after PLR | during one hour , the day of inclusion
  Measure of cardiac output with Physioflow after passive leg raising maneuver (PLR)

SECONDARY OUTCOMES:
Measure of cardiac output with transthoracic echocardiography (TTE) after volume expansion | during one hour , the day of inclusion
  Measure of cardiac output with transthoracic echocardiography (TTE) after volume expansion
Measure of cardiac output with Physioflow after volume expansion | during one hour , the day of inclusion
  Measure of cardiac output with Physioflow after volume expansion

CONTACTS AND LOCATIONS:
Overall Officials: Didier Thevenin, MD, Principal Investigator — Centre Hospitalier de Lens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No